CLINICAL TRIAL: NCT06636513
Title: A Single-arm, Open-label Clinical Trial to Evaluate the Effect of SMT04 in Irritable Bowel Syndrome (IBS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: GenieBiome Limited (Industry); National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Ang Shih Wen Daphne, Senior Consultant, Changi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBSXtra
Record Dates: First submitted 2024-08-20; First posted 2024-10-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: probiotic; IBS; microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: This is a pilot prospective single-arm, open-label clinical trial to assess the effect of the probiotic SMT04 (M3XTRA) on IBS symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SMT04 Arm (Experimental): Each subject will take 1 sachet of SMT04 daily for 3 months.
  Interventions: Dietary Supplement: SMT04 (M3XTRA)

INTERVENTIONS:
Dietary Supplement: SMT04 (M3XTRA) — This is a pilot prospective single-arm, open-label clinical trial to assess the effect of the probiotic SMT04 (M3XTRA) on the gut microbiome and relief of IBS symptoms.

SUMMARY:
Probiotic supplements improve IBS symptoms through manipulation of the gut microbiota. Metabolites derived from microbiota metabolism and host-microbiota co-metabolism have an impact on host intracellular signalling pathways. Although probiotic supplements improve IBS symptoms, the precise composition of probiotics that can achieve optimal response remains unclear. SMT04 (M3XTRA, GenieBiome Limited, Hong Kong, China) is a novel product that is commercially available as a dietary supplement in Singapore. It consists of a patented probiotics blend of 5 probiotics (3 Bifidobacteria and 2 Streptococci with 12.5 billion CFU in 1 sachet). Probiotics preparation that included varying composition of Bifidobacteria and Streptococci strains had previously demonstrated efficacy in achieving symptom improvement in IBS patients. Streptococcus thermophilus, a component of the blended probiotics, significantly improved intestinal functional barrier in healthy subjects. Thus there is potential for SMT04, a dietary supplement, to be a treatment option for IBS patients. This is a multi-centered trial, all data and samples from the study sites will be pooled together for analysis.

DETAILED DESCRIPTION:
Probiotic supplements improve IBS symptoms through manipulation of the gut microbiota. Metabolites derived from microbiota metabolism and host-microbiota co-metabolism have an impact on host intracellular signalling pathways. Although probiotic supplements improve IBS symptoms, the precise composition of probiotics that can achieve optimal response remains unclear. SMT04 (M3XTRA, GenieBiome Limited, Hong Kong, China) is a novel product that is commercially available as a dietary supplement in Singapore. Probiotics preparation that included varying composition of Bifidobacteria and Streptococci strains had previously demonstrated efficacy in achieving symptom improvement in IBS patients. Streptococcus thermophilus, a component of the blended probiotics, significantly improved intestinal functional barrier in healthy subjects. Thus there is potential for SMT04, a dietary supplement, to be a treatment option for IBS patients.

The central hypothesis is that SMT04 can modulate gut microbiota and improve clinical symptoms of subjects with IBS. This pilot study will evaluate the effect of SMT04 on improving IBS related scores and the longitudinal changes in gut microbiome.

The investigators hypothesize that SMT04 can modulate gut microbiota and improve the clinical symptoms of subjects with IBS. This pilot study will examine the effect of SMT04 probiotic supplementation on symptoms in IBS patients. The Rome III rather than Rome IV IBS diagnostic criteria will be used as it is less restrictive with less temporal fluctuation, and hence will be more suitable in an exploratory study. The study will also analyse the longitudinal changes in gut microbiome composition to correlate clinical outcomes with pathophysiological changes. This is a multi-centered trial, all data and samples from the study sites will be pooled together for analysis. If this pilot study demonstrates potential beneficial effect, the investigators will conduct a more definitive randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 21 years to 70 years old
* Meet the criteria of the Rome-III-definition of IBS with diarrhoea or mixed subtypes, or functional diarrhoea Rome-III-definition: Abdominal pain or abdominal discomfort on minimum of three days per month during the last three months, starting at least six months ago, and a minimum of two of the following criteria:

  * Improvement of symptoms after defecation
  * Start of symptoms in association with a change in stool frequency
  * Start of symptoms in association with a change in stool consistency Subtype of IBS-D which requires more than 25% of the participant's stools to be loose and less than 25% hard and lumpy; subtype of IBS-M which the participant's stools must be both hard and lumpy, as well as loose in consistency at least 25% of the time. Functional diarrhoea: The experience of loose or watery stools without pain occurring in at least 75% of bowel movements for at least three months over the last six months.
* Have the latest negative colonoscopy result within five years
* Literate and can complete questionnaire
* Written informed consent is obtained

Exclusion Criteria:

* Known inflammatory bowel disease, lactose intolerance or other malabsorption syndromes, celiac disease, diabetes mellitus, thyroid dysfunction, cancer, immunodeficiency, autoimmune diseases, severe hepatic or renal insufficiency, other explainable causes of abdominal pain, diarrhoea or constipation
* Known operations involving small intestines and large intestines; or history of appendectomy, hysterectomy, and cholecystectomy in last 6 months.
* Known severe mental illnesses; unstable type or dose of psychiatric drugs within the last 3 months that will affect their judgement of study participation.
* Evidence of active infection at the time of inclusion
* History of use of prebiotics, probiotics, antibiotic therapy or anti-inflammatory drugs within the last 2 weeks
* Known current pregnancy or breast-feeding female

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in microbiota (measured using Shannon index, Principal coordinate analysis, heatmaps) at month 3 after taking SMT04 | 3 months
  Assess change in microbiota (alpha diversity, beta diversity, taxonomic abundances) at Month 3

SECONDARY OUTCOMES:
The improvement of irritable bowel syndrome - severity scoring system (IBS-SSS) score at month 3 (Minimal symptoms 0-74; Mild symptoms 75-174; Moderate symptoms 175-299; Severe symptoms 300-500) | 3 months
  Examine improvement of IBS-SSS score at Month 3
Improvement in gastrointestinal symptoms against baseline as measured by GI symptom assessment (improved, unchanged or worsened) | 3 months
  Change in gastrointestinal symptoms (presence/ absence of nausea, vomiting, abdominal pain, bloating, diarrhea, constipation and other symptoms) at Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Shih Wen Ang, Principal Investigator — Changi General Hospital
Locations (1):
- Dr Daphne Ang Shih Wen, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jafari E, Vahedi H, Merat S, Momtahen S, Riahi A. Therapeutic effects, tolerability and safety of a multi-strain probiotic in Iranian adults with irritable bowel syndrome and bloating. Arch Iran Med. 2014 Jul;17(7):466-70. PMID 24979556
- [Background] Mezzasalma V, Manfrini E, Ferri E, Sandionigi A, La Ferla B, Schiano I, Michelotti A, Nobile V, Labra M, Di Gennaro P. A Randomized, Double-Blind, Placebo-Controlled Trial: The Efficacy of Multispecies Probiotic Supplementation in Alleviating Symptoms of Irritable Bowel Syndrome Associated with Constipation. Biomed Res Int. 2016;2016:4740907. doi: 10.1155/2016/4740907. Epub 2016 Aug 9. PMID 27595104